CLINICAL TRIAL: NCT02168920
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Aripiprazole in the Treatment of Patients With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: Aripiprazole for the Treatment of Patients With Agitation Associated With Dementia of the Alzheimer's Type
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It was difficult to secure enrollment of the targeted number of subjects.
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-13-001
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Agitation Associated With Dementia of the Alzheimer's Type
Keywords: Alzeheimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aripiprazole, 2 mg/day (Experimental)
  Interventions: Drug: 2 mg/day
- Aripiprazole, 3 mg/day (Experimental)
  Interventions: Drug: 3 mg/day
- Aripiprazole, 6 mg/day (Experimental)
  Interventions: Drug: 6 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (0 mg/day)

INTERVENTIONS:
Drug: 2 mg/day — Once daily for 10 weeks
  Arms: Aripiprazole, 2 mg/day
Drug: 3 mg/day — Once daily for 10 weeks
  Arms: Aripiprazole, 3 mg/day
Drug: 6 mg/day — Once daily for 10 weeks
  Arms: Aripiprazole, 6 mg/day
Drug: Placebo (0 mg/day) — Once daily for 10 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy (based on mean change in Cohen-Mansfield Agitation Inventory [CMAI] total score from baseline as the primary efficacy variable), dose-response, and safety of aripiprazole at 2, 3, and 6 mg/day in comparison with placebo in patients with agitation associated with Alzheimer's type dementia

DETAILED DESCRIPTION:
This trial is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, comparison trial to assess the efficacy and safety of aripiprazole in patients with agitation associated with Alzheimer's type dementia. Screening period is 4 weeks. Patients are randomly assigned to one of 4 groups, and treatment period is 10 weeks. Period of post-treatment observation is 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose legal representatives can provide informed consent (Informed consent from the patients where possible).
* Patients who satisfy both of the following diagnostic criteria:

  * Diagnosis of major neurocognitive disorder due to Alzheimer's disease according to Diagnostic and Statistical Manual of mental disorders (DSM-5)
  * Diagnosis of probable Alzheimer's disease according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
* Hospitalized patients or care facility patients
* Patients with an Mini-Mental State Examination (MMSE) score of 1 to 22

Exclusion Criteria:

* Patients with complications of dementia or memory impairment other than Alzheimer's type dementia
* Dementia patients with a Modified Hachinski Ischemic Score of 5 or higher
* Patients with psychological symptoms or behavioral disorders that are clearly due to other medical conditions or substances
* Patients with a complication or history of stroke or transient ischemic attack, except for asymptomatic stroke
* Patients with heart failure classified as New York Heart Asscoiation (NYHA） III or IV
* Patients who require drug therapy for arrhythmia or ischemic heart disease
* Body weight of less than 30 kg
* Patients with a high risk of suicide
* Patients with a complication or history of seizure disorder
* Patients with a complication or history of neuroleptic malignant syndrome, tardive dyskinesia, paralytic ileus, or rhabdomyolysis
* Patients with thyroid disease (except if the disease has been stabilized with drug therapy for 3 months or longer prior to time of informed consent)

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

PRIMARY OUTCOMES:
CMAI | Baseline, 10 weeks
  Change from baseline

SECONDARY OUTCOMES:
Clinical Global Impression of Severity （CGI-S） | Baseline, 10 weeks
  Change from baseline
Clinical Global Impression-Improvement (CGI-I) | 10 Weeks
  Score after 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kanto Region, Japan